CLINICAL TRIAL: NCT01313520
Title: A Randomized Clinical Trial to Study the Effects of Infliximab on Clinical Efficacy and Hand and Wrist Magnetic Resonance Imaging (MRI) in Patients With Active Rheumatoid Arthritis (RA)(Protocol No. P08136)
Brief Title: A Study to Evaluate the Effectiveness of Infliximab and Changes in Hand and Wrist Magnetic Resonance Imaging (MRI) in Participants With Active Rheumatoid Arthritis (RA) (P08136)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P08136; 2011-000079-14 (EudraCT Number)
Record Dates: First submitted 2011-02-25; First posted 2011-03-11 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infliximab (Experimental): 3 mg/kg of Infliximab intravenous infusion
  Interventions: Drug: Infliximab
- Placebo (Placebo Comparator): saline via intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Infliximab — 3 mg/kg of Infliximab at Weeks 0, 2, 6, 14 via intravenous infusion
  Other Names: SCH 215596; Remicade
  Arms: Infliximab
Drug: Placebo — 250 mL of 0.9% sodium chloride at Weeks 0, 2, 6, 14 via intravenous infusion
  Arms: Placebo

SUMMARY:
This is a study to compare the effect of infliximab versus placebo on synovial inflammation as measured by dynamic contrast enhanced (DCE)-MRI of one wrist. The primary hypothesis is that over 14 weeks of therapy, the change from baseline in the volume transfer rate in enhancing synovium is larger due to treatment with infliximab than with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical diagnosis of rheumatoid arthritis for at least 6 months
* Must have at least 6 tender joints AND 6 swollen joints
* Has a C-reactive protein ≥ 1.0 mg/L OR Erythrocyte Sedimentation Rate (ESR) ≥ 28 mm/hr
* Baseline MRI must show evidence of synovitis in the wrist
* Must have screening laboratory tests within acceptable levels
* Women of childbearing potential and all men must agree to use a medically accepted method of contraception prior to entering the study and continue throughout study up to 6 weeks after study completion
* Must meet tuberculosis (TB) screening criteria
* Have received methotrexate therapy for ≥ 3 months; dose must be stable for at least 8 weeks
* If taking the a disease modifying anti-rheumatic drug (DMARD) in combination with methotrexate must be on a stable dose
* Must have a clinically acceptable 12 lead electrocardiogram (ECG)
* If taking oral corticosteroids must be on a stable dose equivalent to ≤10 mg of prednisone (or prednisolone) per day for ≥2 weeks
* If taking daily non-steroidal anti-inflammatory drug (NSAID) must be on a stable dose for ≥2 weeks; if taking NSAID on an as-needed basis must agree to discontinue use for at least 3 days and use only acetaminophen for breakthrough pain for 3 days before each MRI and clinic visit
* If received biological therapies, the last dose of these drugs was to be received ≥ 3 months prior to the baseline visit AND the reason for discontinuations was not for safety considerations OR lack of efficacy

Exclusion Criteria:

* Are pregnant, intend to become pregnant, or are breastfeeding
* Has inflammatory arthritis other than RA
* Has uncontrolled hypertension
* Has moderate or severe congestive heart failure
* Has a history of or current signs and/or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, cerebral, or psychiatric disease
* Has a history of demyelinating disease or symptoms suggestive of multiple sclerosis or optic neuritis
* Is currently participating in another clinical study or have participated in a clinical study (e.g., laboratory or clinical evaluation) within 4 weeks
* Has history of any tumor with the exception of adequately treated basal cell carcinoma or carcinoma in situ of the cervix
* Has a history of any latent or active granulomatous infection including histoplasmosis, or coccidiomycosis
* Had a non-tuberculous mycobacterial infection or opportunistic infection (e.g. cytomegalovirus, Pneumocystis carinii, aspergillosis) within 6 months
* Has a history of an infected joint prosthesis which has not been removed or replaced
* Has a known hypersensitivity to human immunoglobulin proteins or other components of infliximab
* Has received rituximab or natalizumab
* Has known claustrophobia or other contraindication to MRI
* Does not meet washout period guidelines for previous treatments/injections/vaccinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2012-03-01 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Beals C, Baumgartner R, Peterfy C, Balanescu A, Mirea G, Harabagiu A, Popa S, Cheng A, Feng D, Ashton E, DiCarlo J, Vallee MH, Dardzinski BJ. Magnetic resonance imaging of the hand and wrist in a randomized, double-blind, multicenter, placebo-controlled trial of infliximab for rheumatoid arthritis: Comparison of dynamic contrast enhanced assessments with semi-quantitative scoring. PLoS One. 2017 Dec 13;12(12):e0187397. doi: 10.1371/journal.pone.0187397. eCollection 2017. PMID 29236711
- [Derived] MacIsaac KD, Baumgartner R, Kang J, Loboda A, Peterfy C, DiCarlo J, Riek J, Beals C. Pre-treatment whole blood gene expression is associated with 14-week response assessed by dynamic contrast enhanced magnetic resonance imaging in infliximab-treated rheumatoid arthritis patients. PLoS One. 2014 Dec 12;9(12):e113937. doi: 10.1371/journal.pone.0113937. eCollection 2014. PMID 25504080

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infliximab | Placebo
Started | 30 | 31
Completed | 30 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab | Placebo | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (9.5) | 50.1 (10.7) | 50.2 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Volume Transfer Rate From the Blood Plasma to the Enhancing Synovium (Ktrans)
Description: Dynamic Contrast Enhanced (DCE) Magnetic Resonance Imaging (MRI) was performed on one hand at baseline, and then at treatment week 14 to measure the rate constant of transfer of contrast (Ktrans).
Time Frame: Baseline and week 14
Population: Participants treated with infliximab or placebo
Measure: Least Squares Mean (95% Confidence Interval); unit: min ^-1
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 31
min ^-1 | -0.2 [-0.3 to -0.1] | 0.1 [-0.0 to 0.2]
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.4 to -0.1]

2. Secondary Outcome: Percentage of Responders With a 20% Improvement From Baseline in American College of Rheumatology (ACR) Responder Criteria for Tender and Swollen Joints (ACR20).
Description: ACR20 requires that both tender and swollen joint counts improve by at least 20% from baseline, as well as a 20% improvement in at least 3 other core measures from the following: pain, patient's and physician's global assessment, physical disability and C-reactive protein (CRP).
Time Frame: Baseline and week 14
Population: Participants treated with Infliximab or Placebo
Measure: Number (90% Confidence Interval); unit: percentage of responders
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 31
percentage of responders | 56.7 [41.9 to 70.4] | 32.3 [20.3 to 47.0]
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Test type: Superiority or Other; p = 0.048, Fisher Exact

3. Secondary Outcome: Percentage of Responders With a 50% Improvement From Baseline in American College of Rheumatology (ACR) Responder Criteria for Tender and Swollen Joints (ACR50).
Description: ACR50 requires that both tender and swollen joint counts improve by at least 50% from baseline, as well as a 50% improvement in at least 3 other core measures from the following: pain, patient's and physician's global assessment, physical disability and CRP.
Time Frame: Baseline and week 14
Population: Participants treated with Infliximab or placebo
Measure: Number (90% Confidence Interval); unit: percentage of responders
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 31
percentage of responders | 20.0 [10.7 to 34.2] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Test type: Superiority or Other; p = 0.011, Fisher Exact

4. Other Pre Specified Outcome: Change From Baseline in DAS28 CRP.
Description: DAS28 CRP is a composite index of the following: number of tender joints (28 joint count), number of swollen joints (28 joint count), GADP on a 100 mm VAS and concentration of serum CRP. Scores can range from 2-10; with higher values corresponding to higher disease activity, and lower values to better outcomes.
Time Frame: Baseline and Week 14
Population: Participants treated with infliximab or placebo
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Infliximab: 3 mg/kg of Infliximab via intravenous infusion
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 31
units on a scale | -1.8 (0.18) [-2.2 to -1.5] | -0.8 (0.18) [-1.2 to -0.4]
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Test type: Superiority or Other; p < 0.0001, Constrained longitudinal data analysis

5. Other Pre Specified Outcome: Change From Baseline in RAMRIS Synovitis.
Description: RAMRIS Synovitis is an ordinal scoring system of hand synovitis that is scored from 0 to 3 in 8 locations. The scores can range from 0 to 24, with higher values corresponding to higher disease activity, and lower values to better outcomes.
Time Frame: Baseline and Week 14
Population: Participants treated with infliximab or placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 31
units on a scale | -2.30 (4.25) [0.64 to 1.55] | 0.24 (1.98)
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Test type: Superiority or Other; p = 0.001, van Elteren test

6. Other Pre Specified Outcome: Change From Baseline in RAMRIS Osteitis.
Description: RAMRIS Osteitis is an ordinal scoring system of hand osteitis that is scored from 0 to 3 in 25 locations. The scores can range from 0 to 75, with higher values corresponding to higher disease activity, and lower values to better outcomes.
Time Frame: Baseline and Week 14
Population: Participants treated with infliximab or placebo. One participant in the placebo group missing a baseline value was not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | -3.10 (5.04) [-2 to -1.5] | 0.48 (3.22) [-1 to -0.5]
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Test type: Superiority or Other; p = 0.0005, van Elteren test

7. Secondary Outcome: Change From Baseline in Standardized Z-scores of Composite Endpoint Consisting of Clinical Disease Activity Measure DAS28 CRP + Ktrans.
Description: Clinical disease activity score (DAS28 CRP) is a composite index of the following: number of tender joints (28 joint count), number of swollen joints (28 joint count), Patient Global Assessment of Disease Status (GADP) on a 100 mm visual analog scale (VAS) and concentration of CRP. Ktrans is the volume transfer rate from the blood plasma to the enhancing synovium. The individual endpoints are standardized using z-scores, then the z-scores are averaged to create a composite endpoint by use of O'Brien's global statistic.
Time Frame: Baseline and Week 14
Population: Participants treated with Infliximab or placebo
Measure: Least Squares Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 31
Z-score | -0.8 (0.3) [-1.3 to -0.3] | 0.8 (0.2) [0.3 to 1.2]
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Test type: Superiority or Other; Effect Size = 1.40, 90% CI 2-sided [0.92 to 1.87]

8. Secondary Outcome: Change From Baseline in Standardized Z-scores of Composite Endpoint Consisting of Clinical Disease Activity Measure DAS28 CRP + Rheumatoid Arthritis MRI Score (RAMRIS) Synovitis + RAMRIS Osteitis.
Description: DAS28 CRP is a composite index of the following: number of tender joints (28 joint count), number of swollen joints (28 joint count), GADP on a 100 mm VAS and concentration of CRP. RAMRIS Synovitis is an ordinal scoring system of hand synovitis that is scored from 0 to 3 in 8 locations, ranging from 0 to 24 total. RAMRIS Osteitis is an ordinal scoring system of hand osteitis that is scored from 0 to 3 in 25 locations, ranging from 0 to 75 total. The individual
  endpoints are standardized using z-scores, then the z-scores are averaged to create a composite endpoint by use of O'Brien's global statistic.
Time Frame: Baseline and Week 14
Population: Participants treated with Infliximab or placebo
Measure: Least Squares Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 31
Z-score | -0.7 (0.3) [-1.3 to -0.2] | 0.8 (0.2) [0.2 to 1.3]
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Test type: Superiority or Other; Effect Size = 1.10, 90% CI 2-sided [0.64 to 1.55]

ADVERSE EVENTS:
Arm/Group | Infliximab | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 8/30 | 8/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=30) | Placebo (N=31)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor has the right to review and comment on publications, abstracts, slides and manuscripts and on the data analysis and presentation.